CLINICAL TRIAL: NCT04269096
Title: Compliance With Laparoscopic Cholecystectomy Care Protocol
Brief Title: Laparoscopic Cholecystectomy Care Protocol
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00066577
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Guideline Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Protocol Compliance — Compliance with the Prisma Health-Upstate Laparoscopic Cholecystectomy Perioperative Protocol

SUMMARY:
The purpose of this study is to determine compliance with the Prisma Health-Upstate Laparoscopic Cholecystectomy Perioperative Protocol.

DETAILED DESCRIPTION:
Evidence based medicine calls for the application of scientific advances to clinical care. In an effort to address the most common complications of a surgical procedure, perioperative protocols have recently been created in an effort to apply best practices consistently and enhance the recovery from surgery. In addition to evaluating the validity of the protocol components themselves, it is valuable to measure compliance with said protocol. Failure to complete the steps of a care pathway may be caused by several reasons, and a study of application of these steps may help future efforts at standardization of care.

The purpose of this study is to determine compliance with the Prisma Health-Upstate Laparoscopic Cholecystectomy Perioperative Protocol.

Hospital inpatient data from patient charts, office charts, and hospital medical data systems of Prisma Health-Upstate System will be used to review the records of all patients age 18-75 years, inpatient and outpatient, who had surgery for choledocolithiasis between January 1, 2016 to April 1, 2017.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 years and 75 years who had surgery for choledocholithiasis at Prisma Health-Upstate.

Exclusion Criteria:

* Patients under 18 years of age and older than 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 years and 75 years who had surgery for choledocolithiasis at Prisma Health-Upstate.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Protocol Compliance | 15 months
  Percent compliance with protocol components

SECONDARY OUTCOMES:
Length of Stay | 15 months
  Post acute care unit length of stay will be measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: William Hand, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Memorial Hospital, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No